CLINICAL TRIAL: NCT04191356
Title: An Observational, Multicentre Study to Evaluate the Feasibility of a Novel Mobile Health Monitoring Platform to Capture Patient-centered Outcomes Measures Among Patients With Heart Failure (HF)
Brief Title: Evaluating Mobile Health Tool Use for Capturing Patient-centered Outcomes Measures in HF Patients
Status: Terminated | Type: Observational
Why Stopped: Collected enough data to support the Endpoints
Sponsor: Biofourmis Singapore Pte Ltd. (Industry)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: CT003
Record Dates: First submitted 2019-11-26; First posted 2019-12-09 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure
Keywords: 6MWT; accelerometer; biosensors; wearable
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart Failure (HF) is a highly prevalent disease that also carries high morbidity and mortality. The Food and Drug Administration (FDA) recognizes the importance of developing patient-centric endpoints that are relevant to patients beyond mortality and hospitalizations.

Although functional status can be objectively measured by peak exercise oxygen consumption, it is difficult and impractical to implement in large clinical studies, especially in an ambulatory real-world setting. Recently, new mobile health technologies have emerged as clinical tools and offer an opportunity to overcome these challenges in measuring functional capacity and recording symptoms.

The goal of this observational study is to evaluate the feasibility of monitoring functional capacity among patients with heart failure (HF) using mobile health monitoring platforms.

Everion® and Apple Watch Series 4 and above will be used for this study. The BiovitalsHF® mobile app can capture patients' key cardiopulmonary physiological parameters, functional capacity (using activity patterns, including guided mobile-based 6MWT, audio recording) and assessment of QoL through validated PROs.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible to be included in the study only if all the following criteria apply:

Subjects has provided informed consent prior to initiation of any study specific activities/procedures.

1. Age more than 21 to less than 85 years at signing of informed consent.
2. Diagnosis of heart failure, defined as requiring pharmacologic treatment for heart failure, with NYHA class I to class III at most recent screening assessment
3. Screening within 30 days after Clinic Visit or hospitalization for heart failure - either as a primary or secondary diagnosis.
4. History of (within the past 6 months) or current use of diuretics.
5. HF patient who is willing to comply with study restrictions including Everion device management (wearing and charging the device), Apple watch Series 4 and above device management (wearing and charging the device) and BiovitalsHF Patient App Management (pairing Everion device and Apple watch Series 4 and above and BiovitalsHF Patient App, and carrying the smartphone for answering questionnaires and data reporting)

Exclusion Criteria

Subjects are excluded from the study if any of the following criteria apply:

Disease Related

1. Acute coronary syndrome (ST-elevation myocardial infarction, non-ST-elevation myocardial infarction, unstable angina) stroke, or transient ischemic attack, major cardiac surgery, percutaneous coronary intervention, or valvuloplasty within the 30 days prior to screening.
2. Uncontrolled hypertension defined as sitting systolic blood pressure (SBP) more than or equal to 180 mm Hg or diastolic BP (DBP)more than or equal to 110 mm Hg.
3. Untreated severe ventricular arrhythmia (e.g., ventricular tachycardia or ventricular fibrillation).
4. Symptomatic bradycardia or second or third-degree heart block without a pacemaker

Other Medical Conditions

1. Malignancy except non-melanoma skin cancers, cervical or breast ductal carcinoma in situ within the last 5 years
2. Hospitalization with any pathology that may meaningfully interfere with functional tolerance, cardiopulmonary capacity or mobility within the 30 days prior to screening.
3. Estimated glomerular filtration rate (eGFR) < 20 mL/min/1.73 m2 or receiving dialysis at screening.

Prior/Concomitant Medication

1. Currently receiving treatment or procedure in another investigational device or drug study.

Other Exclusions

1. Likely to receive during the duration of the study, in the opinion of the investigator, planned revascularization, implantation of ICD or CRT, ventricular assist device, continuous or intermittent inotropic therapy, hospice care, or cardiac transplant.
2. Implantable cardioverter defibrillator or initiation of cardiac resynchronization therapy (CRT) (with/without implantable cardioverter defibrillator) within 30 days prior to enrollment.
3. Recipient of any major organ transplant (e.g. lung, liver, heart, bone marrow, kidney).
4. Less than 4 months prior Interventional Clinical Study participation.
5. Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (e.g. Clinical Outcome Assessments) to the best of the subject and investigator's knowledge.
6. History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
7. Any individuals that are lacking the ability to consent.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 150 eligible subjects will be enrolled into the study. Eligible subjects will include adults with a diagnosis of heart failure (NYHA class I to class III), and screened within 30 days after Clinic Visit or hospitalization for heart failure - either as a primary or secondary diagnosis.
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2020-10-17 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of monitoring functional capacity among patients using mobile health monitoring platform | 8 weeks
  Measurement of correlation between physiology and accelerometer (activity) data/derivatives with:
  * 6MWT
  * Patient-reported KCCQ
  * Lab results

SECONDARY OUTCOMES:
Compliance rate | 8 weeks
  Compliance rate to measure the feasibility of collecting continuous, biometrics data and ePROs using mobile-health monitoring platform
Drop-out rate | 8 weeks
  Drop-out rate to measure the feasibility of collecting continuous, biometrics data and ePROs using mobile-health monitoring platform
Mean time worn/day | 8 weeks
  Mean time worn/day to measure the feasibility of collecting continuous, biometrics data and ePROs using mobile-health monitoring platform
Proportion of time worn that device produces reliable data | 8 weeks
  Proportion of time worn that device produces reliable data to measure the feasibility of collecting continuous, biometrics data and ePROs using mobile-health monitoring platform

OTHER OUTCOMES:
Percentage of patients on HF GDMT | 8 weeks
  Percentage of patients on beta blocker, ACE/ARN/ or ARNI and MRA
Percentage of patients on target dose of HF GDMT | 8 weeks
  Target dose of HF GDMT is according to 2021 Update to the 2017 ACC Expert Consensus Decision Pathway for Optimization of Heart Failure Treatment
Unplanned hospital visits of patients on HF GDMT and target dose of GDMT | 8 weeks
  30-days hospitalization, Clinic visits and ED visits, and its correlation to patients on HF GDMT and target dose of GDMT
Questionnaire for patient experience | 8 weeks
  Questionnaire to evaluate the subjects' experience with the mobile device(s) and mobile health monitoring platform
Association of ECG/Vitals/voice-related biomarker to progression of HF disease | 8 weeks
  Ability to detect changes in ECG/Vitals/voice biomarker, and correlate with functional status and clinical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Maulik Majmudar, M.D., Study Chair — Biofourmis Inc.
Locations (6):
- Mayo Clinic, Jacksonville, Florida, United States
- Singapore (5):
  - National University Hospital, Singapore
  - National Heart Centre Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Changi General Hospital, Singapore
  - Khoo Teck Puat Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campbell RT, Jhund PS, Castagno D, Hawkins NM, Petrie MC, McMurray JJ. What have we learned about patients with heart failure and preserved ejection fraction from DIG-PEF, CHARM-preserved, and I-PRESERVE? J Am Coll Cardiol. 2012 Dec 11;60(23):2349-56. doi: 10.1016/j.jacc.2012.04.064. Epub 2012 Nov 7. PMID 23141494
- [Background] Butler J, Hamo CE, Udelson JE, Pitt B, Yancy C, Shah SJ, Desvigne-Nickens P, Bernstein HS, Clark RL, Depre C, Dinh W, Hamer A, Kay-Mugford P, Kramer F, Lefkowitz M, Lewis K, Maya J, Maybaum S, Patel MJ, Pollack PS, Roessig L, Rotman S, Salsali A, Sims JJ, Senni M, Rosano G, Dunnmon P, Stockbridge N, Anker SD, Zile MR, Gheorghiade M. Exploring New Endpoints for Patients With Heart Failure With Preserved Ejection Fraction. Circ Heart Fail. 2016 Nov;9(11):e003358. doi: 10.1161/CIRCHEARTFAILURE.116.003358. PMID 27756791
- [Background] Palau P, Nunez E, Dominguez E, Sanchis J, Nunez J. Physical therapy in heart failure with preserved ejection fraction: A systematic review. Eur J Prev Cardiol. 2016 Jan;23(1):4-13. doi: 10.1177/2047487314562740. Epub 2014 Dec 8. PMID 25488549
- [Background] Hsieh FY, Bloch DA, Larsen MD. A simple method of sample size calculation for linear and logistic regression. Stat Med. 1998 Jul 30;17(14):1623-34. doi: 10.1002/(sici)1097-0258(19980730)17:143.0.co;2-s. PMID 9699234